CLINICAL TRIAL: NCT07148544
Title: The Effect of the Sedo-Analgesia Protocol Applied to Intensive Care Unit Patients on Patient Outcomes
Acronym: Sedo Analgesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Principal Investigator, Ceylan Kisial, Directör, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CU-SBF-CK-02; TDK-2025-17634 (Other: Çukurova University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-08-09; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Neurosurgical Surgery; Sedo-analgesia; İntensive Care; Nursing Care
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group will receive the clinic's routine sedation-analgesia management plan. Patients will be monitored and their vital signs will be recorded upon admission to the intensive care unit. Medications will be administered according to the physician's orders based on improved treatment and analgesia. The nurse responsible for the patient will administer sedatives based on their own observation/assessment and the physician's order, without any sedation-analgesia protocol. The nurse responsible for the patient will also record all treatments as directed by the physician. During follow-up, data collection tools (RASS, HSF, NVPS, and CPOT) will be used to record patients' pain, anxiety, sedation level, GCS, blood gases, and vital signs twice daily, taking into account non-busy family visits and nursing care hours, between 10:00 and 11:00 and 14:00 and 15:00 (before, during, and 30 minutes after).
  Interventions: Other: control group
- Experimental Group (Other): The experimental group will receive an algorithmic sedoanalgesia protocol led by a nurse, and alarm volume will be adjusted in accordance with WHO recommendations. To ensure the patient understands the concept of daytime, the brightness of the lights in the patient's room will be adjusted only after 10:00 PM, ensuring they do not disrupt treatment and care. The patient's primary nurse will then assess the RASS, NVPS, and CPOT for three days. Based on these assessments, the patient will adjust the medication infusion rate and strive to achieve the target scale value range. During follow-up, the researcher will play music twice daily, between 10:00 AM and 11:00 AM and 2:00 PM and 3:00 PM, taking into account non-busy family visits and nursing care hours. Music will be played using pre-recorded music from selected Musi Cure albums for three days. Music will be played for 30 minutes at 10:00 AM and 2:00 PM. Data will be recorded using data collection tools.
  Interventions: Other: Sedo analgesia protocol

INTERVENTIONS:
Other: Sedo analgesia protocol — Nurse-Controlled Sedo-Analgesia Protocol
  Arms: Experimental Group
Other: control group — The clinic's routine sedation analgesia management plan will be implemented.
  Arms: Control Group

SUMMARY:
Neurosurgical interventions are a leading cause of death and disability in adults, and managing intracranial hypertension in the acute phase is a critical treatment process to prevent secondary brain injury . Among surgical and medical interventions to control intracranial pressure, appropriate sedoanalgesia protocols can provide comfort to patients and directly control intracranial pressure by regulating cerebral metabolism . Appropriate sedoanalgesia has been reported in the literature to reduce cerebral metabolic rate, cerebral blood flow, and cerebral blood volume by resting the brain, and has been observed to improve elevated intracranial pressure. Resting the brain means a decrease in cerebral metabolic rate, allowing it to utilize energy more efficiently . This decrease in the brain's need for blood supply decreases, thereby decreasing cerebral blood flow. This reduction in blood flow can help reduce intracranial pressure, as excessive blood flow and fluid accumulation can lead to elevated intracranial pressure. In this regard, sedoanalgesia applications help patients become more stable and better maintain cerebral perfusion pressure . This can help preserve brain function by ensuring adequate oxygen and nutrients to brain tissue . In this context, sedoanalgesia is an important tool in managing intracranial pressure and can be used strategically to improve brain health.

However, inadequate sedoanalgesia may fail to achieve intended treatment goals, while excessive sedoanalgesia can lead to complications associated with lethal sedation. Therefore, it is important to determine the appropriate sedoanalgesia protocol and continuously monitor patient outcomes (such as vital signs, blood gas parameters, pain, sedation scores, and GCS).

As healthcare professionals, nurses, along with physicians, are the decision-makers and implementers in the sedoanalgesia management of critically ill patients in intensive care, ensuring optimal sedoanalgesia, achieving the desired level of sedoanalgesia, optimizing patient comfort, ensuring patient safety, and maintaining sedoanalgesia when indicated. Therefore, our study was designed to evaluate the impact of the sedoanalgesia protocol applied to intensive care patients, including neurosurgical patients, on patient outcomes and is believed to guide the literature.

Keywords: Neurosurgical surgery, Sedo-analgesia, Intensive care, Nursing care

DETAILED DESCRIPTION:
The study is planned as a randomized controlled intervention study to evaluate the effect of the sedo-analgesia protocol applied to intensive care patients on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Undergoing elective or emergency neurosurgical surgery and admitted to intensive care after surgery,
* Postoperative Glasgow Coma Score 9>GCS <13,
* Requiring mechanical ventilation for at least 24 hours,
* Having a RASS score ≥ -4,
* Are hemodynamically stable,
* Receiving intermittent sedation,
* Patients whose relatives consent to the study will be included in the sample criteria.

Exclusion Criteria:

* Those with alcohol or substance abuse,
* Those with known hearing loss,
* Those diagnosed with brain death,
* Those requiring deep sedation, such as those requiring the administration of muscle relaxants, a body mass index (BMI) > 30, or those with conditions that affect consciousness such as hypercapnia, hyperglycemia, or hypoglycemic coma, or those requiring deep sedation such as pulmonary hypertension,
* Those with cognitive impairment such as epilepsy surgery, Huntington's disease, or frontal lobe or cerebral cortex damage,
* Those with any disease that impairs thermoregulation, such as damage to the hypothalamus, which controls the sleep-wake cycle, or damage to the thalamus, which causes disorders such as impaired brain motor functions,
* Those with quadriplegia,
* Those with a serious pulmonary condition (Chronic Obstructive Pulmonary Disease (COPD), asthma, pneumonia, pulmonary embolism, etc.),
* Those with an allergy to opioids (e.g., fentanyl, remifentanil, sufentanil, morphine),
* Those with severe liver disease and renal dysfunction.
* Psychiatric history (schizophrenia, mania, delirium, cognitive impairment, mental retardation).
* Patients who develop brain damage or complications during the study (such as a GCS < 9 drop, rebleeding, status epilepticus, convulsions, mental status disturbance/delirium, vomiting, tremor, myoclonus) will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient Outcomes Form (HSF) | 1 year, 2 years
  The Patient Information Form consists of eight questions regarding patient information.
  Patient Outcomes Form (HSF): This form was developed by researchers based on a literature review to monitor blood gas parameters, vital signs, pain, medication dosage, GCS, NVPS, CPOT, and RASS levels in patients in the experimental and control groups.
Adult Nonverbal Pain Scale (NVPS | 1 year, 2 years
  Adult Nonverbal Pain Scale (NVPS): This scale was developed to assess pain during painful procedures in patients who cannot communicate verbally. It is an important tool for determining pain levels and developing appropriate treatment and care strategies, especially in patients who cannot express pain.
Intensive Care Pain Observation Scale (CPOT) | 1 year, 2 years
  Intensive Care Pain Observation Scale (CPOT): This scale is used to assess pain in patients in the intensive care unit.
Ricmond Sedation Agitation Scale (RASS | 1 year, 2 years
  Ricmond Sedation Agitation Scale (RASS): This scale is used to determine the sedation and agitation levels of seriously ill patients undergoing mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- TC Adana City Training and Research Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For now, I am thinking of publishing it first in my article and doctoral thesis.